CLINICAL TRIAL: NCT02624440
Title: A Randomized, Open-label Phase III Study of Clarithromycin, Sulfamethoxazole/Trimethoprim or Observation in Combination With Standard Therapy in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Clarithromycin, Sulfamethoxazole/Trimethoprim or Observation in Newly Diagnosed Multiple Myeloma
Acronym: SUTRICA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henrik Gregersen (Other)
Collaborators: Danish Myeloma Study Group (Other)
Responsible Party: Sponsor-Investigator, Henrik Gregersen, Consultant, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DMSG#01/12; 2012-004424-38 (EudraCT Number)
Record Dates: First submitted 2015-12-04; First posted 2015-12-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Myeloma; Infection
Keywords: Multiple Myeloma; Infection; Clarithromycin; Trimethoprim-Sulfamethoxazole Combination
MeSH Terms: conditions — Multiple Myeloma; Infections | interventions — Clarithromycin; Trimethoprim, Sulfamethoxazole Drug Combination; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Clarithromycin (Experimental): p.o. clarithromycin 250 mg twice daily for 180 days
  Interventions: Drug: Standard myeloma treatment; Drug: Clarithromycin
- Sulfamethoxazole/trimethoprim (Experimental): p.o. sulfamethoxazole/trimethoprim 400/80 mg twice daily for 180 days
  Interventions: Drug: Standard myeloma treatment; Drug: Sulfamethoxazole/trimethoprim
- Observation (Experimental): Observation without prophylactic antibiotic treatment
  Interventions: Drug: Standard myeloma treatment; Drug: Observation

INTERVENTIONS:
Drug: Standard myeloma treatment — The choice of myeloma standard treatment is at the discretion of the treating investigator guided by the national Danish guidelines for treatment of multiple myeloma
Drug: Clarithromycin — P.o. clarithromycin 250 mg twice daily
  Arms: Clarithromycin
Drug: Sulfamethoxazole/trimethoprim — P.o. sulfamethoxazole/trimethoprim 400/80 mg twice daily
  Arms: Sulfamethoxazole/trimethoprim
Drug: Observation — Observation without prophylactic antibiotic
  Arms: Observation

SUMMARY:
This study evaluates the effect of prophylactic antibiotics in multiple myeloma. One third of patients will received treatment with clarithromycin, one third of patients will receive treatment with sulfamethoxazole/trimethoprim and one third will be observed without prophylactic antibiotics. All patients receive concurrent anti-myeloma treatment.

DETAILED DESCRIPTION:
There is a need for improvement of the prognosis in elderly myeloma patients. The patients are fragile due to age and severe comorbidity. Infections are frequent during the course of initial myeloma treatment and contribute to the high morbidity and mortality in elderly patients. Furthermore infections often lead to delay in myeloma treatment and to dose reduction. The use of primary antibiotic prophylaxis might influence the frequency of these complications. In the study myeloma patients who are ineligible for high-dose melphalan with stem cell support are randomised to either p.o. clarithromycin 250 mg twice daily for 180 days, p.o. sulfamethoxazole/trimethoprim 400/80 mg twice daily for 180 days or observation without prophylactic antibiotics. All patients receive concurrent myeloma treatment at the discretion of the treating physician. The choice of anti-myeloma treatment has to be settled before randomization. The study evaluates the frequency of infections in patients treated with clarithromycin, sulfamethoxazole/trimethoprim or observation

ELIGIBILITY:
Inclusion Criteria:

* Myeloma diagnosis according to IMWG criteria
* Treatment demanding disease
* Signed informed consent given prior to any study related activities, except bone marrow samples for diagnosis, FISH, biobanking, and skeletal x-ray
* Age > 18 years

Exclusion Criteria:

* Allogeneic transplantation scheduled as a part of the treatment
* High-dose melphalan with stem cell support scheduled as a part of the treatment
* Myeloma treatment prior to entry in the study, except radiotherapy, bisphosphonates/denusumab or corticosteroids for symptom control
* Concurrent disease making clarithromycin or sulfamethoxazole/trimethoprim treatment unsuitable
* Positive pregnancy test (only applicable for women with childbearing potential)
* Known or suspected hypersensitivity or intolerance to claritromycin, sulfamethoxazole or trimethoprim
* Prolonged QT corrected (QTc) interval ( > 500 msec on screening ECG)
* Concurrent treatment with cabergoline, fluconazole, ketoconazole, pimozide, quetiapine, sirolimus, verapamil, tacrolimus, ergot alkaloid or methotrexate
* Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrolment, uncontrolled angina or known cardiac amyloidosis
* Severe renal dysfunction (estimated creatinine clearance <10 mL/min)
* Serious medical or psychiatric illness which, in the judgment of the investigator, would make the patient inappropriate for entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of frequency of infections in patients treated with clarithromycin, sulfamethoxazole/trimethoprim or observed without prophylactic antibiotic | One year

SECONDARY OUTCOMES:
Response rates in the group of patients treated with clarithromycin compared to the other patients in the study | One year
Comparison of adverse events assessed by CTCAE v4.0 in patients treated with clarithromycin, sulfamethoxazole/trimethoprim or observed without prophylactic antibiotic | 6 months
Comparison of overall survival between patients treated with clarithromycin, sulfamethoxazole/trimethoprim or observed without prophylactic antibiotic | Three years
Quality of life assessed by EORTC QLQ-MY20 | One year
Quality of life assessed by EORTC QLQ-C30 | One year

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Gregersen, MD, Principal Investigator — Aalborg University Hospital
Locations (8):
- Denmark (8):
  - Department of Hematology, Aalborg University Hospital, Aalborg
  - Department of Hematology, Aarhus University Hospital, Aarhus
  - Department of Hematology, Rigshospitalet, Copenhagen
  - Department of Hematology, Esbjerg Sygehus, Esbjerg
  - Department of Hematology, Herlev Hospital, Herlev
  - Department of Hematology, Hospitalsenheden Vest, Holstebro
  - Department of Hematology, Odense University Hospital, Odense
  - Department of Hematology, Roskilde Hospital, Roskilde